CLINICAL TRIAL: NCT03928665
Title: Long-term Observation of Ophthalmic Changes in Patients With Obstructive Sleep Apnea
Status: Active, not recruiting | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Collaborators: Wrocław University of Science and Technology (Other)
Responsible Party: Principal Investigator, Joanna Przeździecka-Dołyk, Investigator, Wroclaw Medical University
Other Study IDs: ST.2012.001
Record Dates: First submitted 2019-04-14; First posted 2019-04-26 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Sleep Apnea; Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Sleep Apnea Syndromes; Glaucoma; Ocular Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control group
- Sleep apnea using CEPAP
- Sleep apnea not using CEPAP
- Glaucoma control group

SUMMARY:
The ophthalmic changes during long-lasting sleep apnea are lacking in description and assessment. The investigators intend to observe patients for a long time and observe if the changes in eye tissues are progressing over the years in easily recognizable patterns.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed obstructive sleep apnea indicated for positive airway pressure therapy,
* ongoing treatment of sleep apnea with positive airway pressure therapy,
* patients older than 18 years,
* signed inform consent

Exclusion Criteria:

* pregnant and breastfeeding persons

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult individuals with an indication for therapy with positive airway pressure.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-10-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Perimetry changes over the years | 10 years
  Changes in retinal sensitivity (measured in decibels/ dB) during observation time measured by standard automated perimetry. The manner of presentation of overall descriptors auch as: mean deviation (MD; dB) and pattern standard deviation (PSD; dB) will be recorded.
Flicker defined form perimetry changes over the years | 10 years
  Changes in retinal sensitivity (measured in decibels/ dB) during observation time measured by standard automated perimetry with flicker defined form signal. The manner of presentation of overall descriptors auch as: mean deviation (MD; dB) and pattern standard deviation (PSD; dB) will be recorded.
RareBit perimetry changes over the years | 10 years
  Changes in Changes in retinal sensitivity (measured in percentage of all presented excitors/ %) during observation time measured by RareBit signal perimetry. The manner of presentation of overall descriptors auch as: mean hit rate (MHR; %), area under 90% (%) and sectorial mean miss rate (MMR; %) will be recorded.

SECONDARY OUTCOMES:
Functional Outcomes of Sleep Questionnaire | 10 years
  Quality assessed with the Functional Outcomes of Sleep Questionnaire (FOSQ) comparing the score at baseline with during 10 years of observation. The questionnaire are composed of 30 questions that can be answered from 1 to 4 points (where 1 means extreme difficulty of doing an activity and 4 - no difficulties). Five subscales are given such as: General Productivity (8 questions -1 - 4, 8 - 11), Social Outcome (2 questions - 12, 13), Activity Level (9 questions - 5, 14 - 16, 22 - 26), Vigilance (7 questions - 6, 7, 17 - 21), Intimate Relationships and Sexual Activity (4 questions - 27 - 30). To obtain a Total Score: Calculate the mean of the subscale scores and multiply that mean by the number of subscales for which there is a score. The potential range of scores for the Total Score is 5 - 20.
Epworth Sleepiness Scale | 10 years
  Quality assessed with the Epworth Sleepiness Scale comparing the score at baseline with during 10 years of observation. The questionnaire are composed of 8 questions describing activities during which patient can feel sleepy, each scored from 0 (zero probability to falling asleep) to 3 (very likely that patient will fall asleep).
Pittsburgh Sleep Quality Index | 10 years
  Quality assessed with the Pittsburgh Sleep Quality Index comparing the score at baseline with during 10 years of observation. The questionnaire are composed of 10 questions composed in seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Change in thickness of the retinal nerve fibre layer (RNFL) | 10 years
  A difference in thickness of the retinal nerve fibre layer during the observation time frame.
Change in the optic nerve morphology - standard chart of HRT | 10 years
  A difference in morphology parameters given by HRT (additional information given in supplementary materials) during the observation time frame.
AREDS 2008 Clinical Lens Opacity Grading Procedure | 10 years
  Using AREDS system for classifying cataracts from photographs: AREDS Report No. 4 the lens opacity will be graded. The change in grading during the observation time frame.
Macular changes in optical coherent tomography (OCT) | 10 years
  Evaluation of macular appearance based on the OCT scans. Any changes from normal appearance will be recorded and evaluated.
Disc damage likelihood scale (DDLS) | 10 years
  Evaluation disc damage likelihood scale based on the fundus photographs (based on the visual scale given in additional documents)

OTHER OUTCOMES:
Influence of fogging lens on retinal sensitivity to given trigger (Goldman III) on standard automated and RareBit perimetry | 1 day
  A fogging lens will be applied (a modified by the author protocol of fogging - increasing of +0.5D lens to obtain the reduction in logMAR visual acuity by 0.2 from best-corrected visual acuity/ BCVA)
Influence of tiredness on retinal sensitivity to given trigger (Goldman III) on standard automated and RareBit perimetry | 1 day
  Influence of different examinations that precedes visual field examination on the perimetry test results (MD and PSD, or MHR, MMR and area under 90%).
Peripapillar and macular vessels density | 5 years
  Measured on the custom-derived protocol and manufacturer software macular and peripapillar vessels density - Angio OCT (OCTA)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Misiuk-Hojło, Professor, Study Chair — Wrocław Medical University
Locations (1):
- Department of Ophthalmology, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chasens ER, Ratcliffe SJ, Weaver TE. Development of the FOSQ-10: a short version of the Functional Outcomes of Sleep Questionnaire. Sleep. 2009 Jul;32(7):915-9. doi: 10.1093/sleep/32.7.915. PMID 19639754
- [Background] Oddone F, Centofanti M, Rossetti L, Iester M, Fogagnolo P, Capris E, Manni G. Exploring the Heidelberg Retinal Tomograph 3 diagnostic accuracy across disc sizes and glaucoma stages: a multicenter study. Ophthalmology. 2008 Aug;115(8):1358-65, 1365.e1-3. doi: 10.1016/j.ophtha.2008.01.007. Epub 2008 Mar 5. PMID 18321579
- Available data/document: DDLS - reference — https://www.sign.ac.uk/assets/sign144_disc_chart_colour.pdf